CLINICAL TRIAL: NCT05753371
Title: Bioequivalence Study of Metformin Hydrochloride 500 mg Film-Coated Tablets in Indonesia Healthy Subject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Pyridam Farma Tbk (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 634/STD/PML/2021
Record Dates: First submitted 2023-02-12; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Drug Use
Keywords: Metformin hydrochloride 500 mg; Bioequivalence study; Pharmacokinetics; Indonesian healthy subject
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glufor® 500 mg film-coated tablet (Experimental)
  Interventions: Drug: Metformin Hydrochloride 500 MG
- Glucophage® 500 mg film-coated tablet (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride 500 MG

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — Metformin is an antihyperglycemic drug used in the management of type-2 diabetes. Metformin hydrochloride improves glucose tolerance in patients with type 2 diabetes, lowering both basal and postprandial plasma glucose. Metformin decreases hepatic glucose production, decreases intestinal absorption of glucose and improves insulin sensitivity by increasing peripheral glucose uptake and utilization.

SUMMARY:
The objective of this present study was to investigate whether Glufor® 500 (metformin hydrochloride 500 mg) film-coated tablets manufactured by PT. Pyridam Farma Tbk is bioequivalent to its reference product, Glucophage® 500 mg film-coated tablets manufactured by PT. Merck Tbk, Indonesia under licensed Merck Sante SAS, France.

DETAILED DESCRIPTION:
Twenty-four subjects were given a single dose of 500 mg Metformin film-coated tablet of either formulation (test or reference) with 240 mL of a 20% glucose solution in water.

ELIGIBILITY:
The inclusion criterias were healthy male or female subjects who/with:

* had read the subject information and signed informed consent documents
* age range from 18 - 55 years
* body mass index between 18 - 25 kg/m2
* had a normal electrocardiogram
* had the blood pressure within normal range (systolic 90-120 mmHg and diastolic 60-80 mmHg)
* had the heart rate within normal range (60 - 100 bpm)
* had absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening.

Exclusion criterias

The subjects' exclusion criterias for the study were:

* those who were pregnant and/or nursing women.
* those with history of contraindication or hypersensitivity to metformin or other antidiabetic agent or other ingredients in the study products or a history of serious allergic reaction to any drug, a significant allergic disease, or allergic reaction.
* those with a history or presence of medical condition which might significantly influence the pharmacokinetic of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.
* those with a history or presence of any coagulation disorder or clinically significant hematology abnormalities.
* those who were using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day.
* those who had participated in any clinical study within 3 months prior to the study (<90 days).
* those who had donated or lost 300 ml (or more) of blood within 3 months prior to the study.
* those who smoked more than 10 cigarettes a day
* those with a history of travelling to another city within the last 14 days
* those with a history of direct contact with a COVID-19 positive person in the subject's neighbourhood
* those with a history or present of sore throat, fever (with temperature more than 37°C) or dyspnea with in the last 14 days
* those who are positive to SARS CoV-2 antigen test
* those who were positive to HIV, HBsAg, and HCV tests (to be kept confidential).
* those with a history of drug or alcohol abuse within 12 months prior to screening for this study.
* those who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access.

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio | 0-24 hours post dose
  The ratio between maximum concentration of test drug and reference drug after drug administration
Geometric Mean Ratio | 0-24 hours post dose
  The ratio between area under curve from 0 to 24 hours of test drug and reference drug

SECONDARY OUTCOMES:
Pharmacokinetics Parameter | 0-24 hours post dose
  Maximum plasma concentration (Cmax)
Pharmacokinetics Parameter | 0-24 hours post dose
  Area Under Curve from 0 to 24 hours (AUCt)

CONTACTS AND LOCATIONS:
Overall Officials: Frans D Suyatna, Principal Investigator — PT Pharma Metric Labs; I Gusti Putu Bagus Diana Virgo, Study Director — PT Pharma Metric Labs
Locations (1):
- PT Pharma Metric Labs, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Al Hawari S, AlGaai E, Yusuf A, Abdelgaleel A, Hammami MM. Bioequivalence study of two metformin formulations. Arzneimittelforschung. 2007;57(4):192-5. doi: 10.1055/s-0031-1296605. PMID 17515289
- [Background] Batolar LS, Iqbal M, Monif T, Khuroo A, Sharma PL. Bioequivalence and pharmacokinetic comparison of 3 metformin extended/sustained release tablets in healthy Indian male volunteers. Arzneimittelforschung. 2012 Jan;62(1):22-6. doi: 10.1055/s-0031-1295428. Epub 2012 Jan 10. PMID 22331759
- See also: Related Info — https://www.accessdata.fda.gov/drugsatfda_docs/psg/Metformin_HCl_ERtab_21574_RC3-09.pdf
- See also: Related Info — https://asean.org/wp-content/uploads/2012/10/BE_Guideline_FinalMarch2015_endorsed_22PPWG.pdf